CLINICAL TRIAL: NCT00889226
Title: A Randomized, Open Label, Dose Titration Study to Evaluate the Efficacy and Safety of Pitavastatin Compared to atoRvastatin in Type 2 dIabeTes Mellitus With Hypercholesterolemia
Brief Title: Efficacy and Safety Study of Pitavastatin Compared to atoRvastatin in Type 2 dIabeTes Mellitus With Hypercholesterolemia
Acronym: ESPRIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWP_PTV4_704
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-07

CONDITIONS: Hypercholesterolemia With Type2DM
Keywords: pitavastatin; PWV; ESPRIT; Pitavastatin and Atorvastatin; Adiponectin; fasting insulin; hs-CRP; baPWV
MeSH Terms: interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitavastatin Group (Experimental)
  Interventions: Drug: Pitavastatin
- Atorvastatin Group (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — Drug: Pitavastatin 2mg daily for 8wks after initial visit. After assessment of LDL-C <100mg/dL at 8wks → Dose adjustment Yes → 2mg daily for second 8wks No → 4mg daily for second 8wks
  Other Names: Livalo
  Arms: Pitavastatin Group
Drug: Atorvastatin — Drug: Atorvastatin 10mg daily for 8wks after initial visit. After assessment of LDL-C <100mg/dL at 8wks → Dose adjustment Yes → 10mg daily for second 8wks No → 20mg daily for second 8wks
  Other Names: Lipitor
  Arms: Atorvastatin Group

SUMMARY:
A randomized, open label, dose titration study to evaluate the efficacy and safety of Pitavastatin compared to atorvastatin in Type 2 Diabetes Mellitus with hypercholesterolemia

DETAILED DESCRIPTION:
To evaluate the effect of pitavastatin compared to atorvastatin on the change of Lipid profiles, ApoA1, ApoB, adiponectin and baPWV as a marker of atherosclerosis in Type 2DM .

ELIGIBILITY:
Inclusion Criteria:

* Age: 25yrs~75yrs
* Fasting TG <400mg/dL, LDL-C ≥130mg/dL
* 3months > Diagnosed Type2 DM, With OAD, HbA1c ≤ 10.0% or First Diagnosed Type2 DM, 6.5%≤HbA1c≤10.0%

Exclusion Criteria:

* Type1 DM, Gestational diabetes
* Patient need to treat with Insulin
* Patient with operational treatment for severe diabetic complication
* Uncontrolled Hypothyroidism
* Unstable angina, MI, transient ischemic attack(TIA), Stroke, PCI, Heart Failure within 3 months (NYHA class4)
* Severe Hypertension (SBP ≥ 180 or DBP ≥ 110mmHg)
* Renal disorder (Serum creatinine ≥ 2.0mg/dL)
* Hepatic disorder (AST or ALT ≥ 2.5 X UNL)
* Creatinine Kinase > 2.5 X UNL
* Gravida or lactation phase
* Administration of Atorvastatin, Rosuvastatin, Pitavastatin

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ho Young Shon, MD, Principal Investigator — Endocrinology, Kangnam Saint Mary's Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pitavastatin Group | Atorvastatin Group
Started | 83 | 78
Completed | 58 | 43
Not Completed | 25 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin Group | Atorvastatin Group | Total
Number analyzed (Participants) | 83 | 78 | 161
Age, Continuous [Mean (Full Range); unit: years] | 59.6 [35.0 to 74.0] | 59.1 [41.0 to 74.0] | 59.3 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 28 | 24 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 83 | 78 | 161

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving LDL- C<100mg/dL
Description: compare the proportion of patients achieving LDL- C<100mg/dL
Time Frame: After 16wk drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Pitavastatin Group | Atorvastatin Group
Number analyzed (Participants) | 80 | 68
Participants | 61 | 54

2. Secondary Outcome: The Change of LDL-C
Description: The change of LDL-C between at 16-week and baseline
Time Frame: After 16wk drug administration
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Pitavastatin Group | Atorvastatin Group
Number analyzed (Participants) | 80 | 68
mg/dl | -69.8 (22.5) | -70.9 (28.2)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Pitavastatin Group | Atorvastatin Group
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/70
Other Adverse Events (participants affected / at risk) | 3/81 | 0/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pitavastatin Group (N=81) | Atorvastatin Group (N=70)
coughing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No